CLINICAL TRIAL: NCT05378113
Title: Ondansetron As a Strategy for Reducing Propofol Injection Pain in Pediatrics: a Randomized Controlled Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, VBansal, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00001599
Record Dates: First submitted 2022-05-12; First posted 2022-05-18 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Injection Site Irritation
Keywords: Injection site pain; Propofol; Ondansetron
MeSH Terms: interventions — Ondansetron; Lidocaine; Injections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ondansetron premedication Group (Experimental): The ondansetron group will receive ondansetron 0.15mg/kg IV push followed immediately by propofol 2mg/kg IV for induction. A 10cc normal saline flush will follow injection of propofol.
  Interventions: Drug: Ondansetron
- Lidocaine premedication Group (Active Comparator): The lidocaine group will receive lidocaine 2% 1mg/kg IV push followed immediately by propofol 2mg/kg IV for induction. A 10cc normal saline flush will follow injection of propofol.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Ondansetron — Ondansetron (Zofran) is a 5-hydroxytryptamine-3 (5-HT3) receptor antagonist commonly used to treat postoperative nausea and vomiting.
  Other Names: Zofran, Ondansetron hydrochloride
  Arms: Ondansetron premedication Group
Drug: Lidocaine — Lidocaine is a local anesthetic agent used intravenously prior to the propofol injection. Currently the standard of care to help decrease the severity of pain in the injection site, a common side effect of propofol.
  Other Names: Xylocaine, lidocaine hydrochloride (HCl) Injection
  Arms: Lidocaine premedication Group

SUMMARY:
This study is a randomized, single-site clinical trial that will take place at Children's Healthcare of Atlanta at Egleston. The investigators want to see if in pediatric patients, giving Zofran prior to propofol, reduces the pain that patients often experience when propofol is injected through an IV. Subjects will be randomized to 1 of 2 groups: lidocaine (common standard of care), or Zofran. The investigators hope to show a means of improving pain control in their patients undergoing anesthesia.

DETAILED DESCRIPTION:
Propofol is a drug commonly used at the beginning of anesthesia (induction). Patients often experience discomfort when propofol is injected through an IV. Ondansetron (Zofran) is a drug that is commonly used to treat nausea after anesthesia. In adult studies, it has been shown that there is significantly less pain when Zofran is given just before propofol is given. The investigators want to see if giving Zofran prior to propofol reduces the pain and discomfort experienced by pediatric patients.

This study is a randomized, single-site clinical trial that will take place at Children's Healthcare of Atlanta at Egleston. Subjects will be randomized to 1 of 2 groups: lidocaine (common standard of care), or Zofran. During induction the treating anesthesiologist will be blinded to the study arm, however they will be unblinded at the end of induction. All subjects will receive Zofran at some point during the surgery - for patients not in the Zofran arm, they will receive it at the end of the case as usual. A blinded observer will score the subject's pain during propofol injection and vital signs will be recorded.

Subjects will be identified by the study team from the surgery schedule. Patients ages 2-17 undergoing surgery with peripheral vascular access (an IV) will be approached. Consent and assent (when appropriate) will be obtained. Subjects will not be compensated. Participation will consist only of the single duration of the surgery.

In this study the investigators hope to show a means of improving pain control in their patients undergoing anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients 2 years old through 17 years of age
* Children undergoing surgery at Children's Healthcare of Atlanta Egleston location
* Patient with existing peripheral vascular access in the arm below the antecubital fossa
* Patients with an American Society of Anesthesiologists (ASA) physical status category score of 1, 2 or 3
* Parent or legal guardian willing to participate, and able to understand and sign the provided informed consent
* No known chronic pain syndrome

Exclusion Criteria:

* Parent or legal guardian unwilling to participate or unable to understand and sign the provided informed consent
* Patients presenting for endoscopy procedures
* Known chronic pain syndrome
* Patient diagnosed with long QT syndrome
* Patient weighing >40kg
* Documented allergy to study medications
* Pain on injection of pre-operative normal saline flush
* Patient has received an opioid within 30 minutes prior to anesthesia induction

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2023-05-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in verbal rating scale (VRS) form baseline | Baseline, during propofol injection (30 seconds)
  Difference in total VRS between the lidocaine and ondansetron groups. Possible score ranges from 0 to 3 with higher scores correlating with worse pain.
Change in Motor score scale from baseline | Baseline, during propofol injection (30 seconds)
  Change in Motor score between the lidocaine and ondansetron groups. Possible score ranges from 0 to 3 with higher scores correlating with worse pain.

CONTACTS AND LOCATIONS:
Overall Officials: Vipin Bansal, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No